CLINICAL TRIAL: NCT07176754
Title: TNF-a Antagonists Attenuate the Systemic Inflammatory Response in Post-cardiac Arrest Syndrome: a Multi Centre, Double-blind, Randomised Controlled Clinical Study
Brief Title: TNF-α Antagonists Mitigate Systemic Inflammatory Response After Cardiac Arrest.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Collaborators: Peking University First Hospital (Other); Peking University People's Hospital (Other); Peking University Shenzhen Hospital (Other); Qilu Hospital of Shandong University (Other); Jiangsu Provincial People's Hospital (Other); Hunan Provincial People's Hospital (Other); Sichuan Provincial People's Hospital (Other); People's Hospital of Guangxi Zhuang Autonomous Region (Other); People's Hospital of Xinjiang Uygur Autonomous Region (Other); Renmin Hospital of Wuhan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00006761-M20250549
Record Dates: First submitted 2025-07-04; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-06

CONDITIONS: Cardiac Arrest (CA); Post Cardiac Arrest Syndrome
Keywords: cardiac arrest; post cardiac arrest syndrome; TNF-α antagonism
MeSH Terms: conditions — Heart Arrest; Post-Cardiac Arrest Syndrome | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Experimental): Patients in the intervention group received a TNF-α antagonist (infliximab) within 6 hours after return of spontaneous circulation(ROSC).
  Interventions: Drug: Infliximab
- control group (Placebo Comparator): Patients in the control group received 250 mL of 0.9% sodium chloride injection as a placebo.
  Interventions: Drug: Sodium chloride injection USP, 0.9% (placebo)

INTERVENTIONS:
Drug: Infliximab — The TNF-α antagonist (infliximab) used by the experimenter was manufactured by Hisun Biopharmaceuticals Ltd. under the trade name "anbaite".The dosage was administered at 5 mg/kg, dissolved in 250 mL of 0.9% sodium chloride injection, and delivered via intravenous infusion over 2 hours.
  Arms: intervention group
Drug: Sodium chloride injection USP, 0.9% (placebo) — Patients in the control group received 250 mL of 0.9% sodium chloride injection as a placebo, administered via intravenous infusion over 2 hours.
  Arms: control group

SUMMARY:
The investigators assessed the effect of TNF-α antagonism within 6 hours of return of spontaneous circulation on 30-day mortality in patients who remained comatose after cardiopulmonary resuscitation (CPR) following cardiac arrest . In addition, the investigators explored the role of this treatment in modulating the systemic inflammatory response and its potential impact on 90- and 180-day morbidity and mortality and neurological outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 years;
2. Patients with suspected cardiogenic cardiac arrest;
3. Patients with comatose state after ROSC (Glasgow Coma Scale [GCS] score <9);
4. Patients with Return of spontaneous circulation (ROSC) sustained for >20 minutes;

Exclusion Criteria:

1. Cardiac arrest due to trauma;
2. Suspected or confirmed hemorrhagic or ischemic stroke;
3. Pregnancy;
4. Cardiac arrest without witnessed collapse;
5. Admission body temperature <30°C;
6. Persistent cardiogenic shock (defined as systolic blood pressure <90 mmHg despite aggressive intervention during screening);
7. Any underlying disease with an expected survival of <180 days;
8. Pre-existing severe neurological dysfunction before cardiac arrest (e.g., Cerebral Performance Category [CPC] 3-4);
9. Time from ROSC to randomization exceeding 4 hours;
10. Left ventricular ejection fraction (LVEF) <35% after ROSC;
11. Known hypersensitivity to TNF-α antagonist components;
12. Known tuberculosis or other active infections;
13. Known poor prognosis (as determined by the investigator);
14. History of liver cirrhosis;
15. History of chronic heart failure with NYHA functional class III-IV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
30-day survival rate | 30 days after randomization.
  All-cause survival rate of patients on day 30 after randomization.

SECONDARY OUTCOMES:
Rate of good neurological function assessed by Modified Rankin scale neurologic function scores and cerebral performance category scores | 30 days, 3 months, and 6 months after randomization
  Modified Rankin scale neurologic function scores and cerebral performance category(CPC) scores at 30 days, 3 months, and 6 months after randomization. Neurological function was assessed using the CPC and mRS scales, with CPC 1-2 and mRS 0-3 scores indicating a good neurological prognosis, and CPC 3-5 and mRS 4-6 scores indicating a poor neurological prognosis.
prolong follow-up survival rate | 3 months and 6 months after randomization
  survival rate
systematic scoring | 24 hours (h), 48 hours, 72 hours and 1 week after randomization
  SOFA score at 24h, 48h, 72h and 1 week after randomization

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Zhou Y, Fan R, Botchway BOA, Zhang Y, Liu X. Infliximab Can Improve Traumatic Brain Injury by Suppressing the Tumor Necrosis Factor Alpha Pathway. Mol Neurobiol. 2021 Jun;58(6):2803-2811. doi: 10.1007/s12035-021-02293-1. Epub 2021 Jan 27. PMID 33501626
- [Result] Chen AQ, Fang Z, Chen XL, Yang S, Zhou YF, Mao L, Xia YP, Jin HJ, Li YN, You MF, Wang XX, Lei H, He QW, Hu B. Microglia-derived TNF-alpha mediates endothelial necroptosis aggravating blood brain-barrier disruption after ischemic stroke. Cell Death Dis. 2019 Jun 20;10(7):487. doi: 10.1038/s41419-019-1716-9. PMID 31221990
- [Result] Yin Z, Raj D, Saiepour N, Van Dam D, Brouwer N, Holtman IR, Eggen BJL, Moller T, Tamm JA, Abdourahman A, Hol EM, Kamphuis W, Bayer TA, De Deyn PP, Boddeke E. Immune hyperreactivity of Abeta plaque-associated microglia in Alzheimer's disease. Neurobiol Aging. 2017 Jul;55:115-122. doi: 10.1016/j.neurobiolaging.2017.03.021. Epub 2017 Mar 27. PMID 28434692
- [Result] Cain BS, Meldrum DR, Dinarello CA, Meng X, Joo KS, Banerjee A, Harken AH. Tumor necrosis factor-alpha and interleukin-1beta synergistically depress human myocardial function. Crit Care Med. 1999 Jul;27(7):1309-18. doi: 10.1097/00003246-199907000-00018. PMID 10446825
- [Result] Stellwagen D, Beattie EC, Seo JY, Malenka RC. Differential regulation of AMPA receptor and GABA receptor trafficking by tumor necrosis factor-alpha. J Neurosci. 2005 Mar 23;25(12):3219-28. doi: 10.1523/JNEUROSCI.4486-04.2005. PMID 15788779
- [Result] Robertson J, Beaulieu JM, Doroudchi MM, Durham HD, Julien JP, Mushynski WE. Apoptotic death of neurons exhibiting peripherin aggregates is mediated by the proinflammatory cytokine tumor necrosis factor-alpha. J Cell Biol. 2001 Oct 15;155(2):217-26. doi: 10.1083/jcb.200107058. Epub 2001 Oct 15. PMID 11604419
- [Result] Lu D, Goussev A, Chen J, Pannu P, Li Y, Mahmood A, Chopp M. Atorvastatin reduces neurological deficit and increases synaptogenesis, angiogenesis, and neuronal survival in rats subjected to traumatic brain injury. J Neurotrauma. 2004 Jan;21(1):21-32. doi: 10.1089/089771504772695913. PMID 14987462
- [Result] Aloisi F, Care A, Borsellino G, Gallo P, Rosa S, Bassani A, Cabibbo A, Testa U, Levi G, Peschle C. Production of hemolymphopoietic cytokines (IL-6, IL-8, colony-stimulating factors) by normal human astrocytes in response to IL-1 beta and tumor necrosis factor-alpha. J Immunol. 1992 Oct 1;149(7):2358-66. PMID 1382099
- [Result] Annborn M, Dankiewicz J, Erlinge D, Hertel S, Rundgren M, Smith JG, Struck J, Friberg H. Procalcitonin after cardiac arrest - an indicator of severity of illness, ischemia-reperfusion injury and outcome. Resuscitation. 2013 Jun;84(6):782-7. doi: 10.1016/j.resuscitation.2013.01.004. Epub 2013 Jan 8. PMID 23313427
- [Result] Tae HJ, Kang IJ, Lee TK, Cho JH, Lee JC, Shin MC, Kim YS, Cho JH, Kim JD, Ahn JH, Park JH, Kim IS, Lee HA, Kim YH, Won MH, Lee YJ. Neuronal injury and tumor necrosis factor-alpha immunoreactivity in the rat hippocampus in the early period of asphyxia-induced cardiac arrest under normothermia. Neural Regen Res. 2017 Dec;12(12):2007-2013. doi: 10.4103/1673-5374.221157. PMID 29323039
- [Result] Nolan JP, Neumar RW, Adrie C, Aibiki M, Berg RA, Bottiger BW, Callaway C, Clark RS, Geocadin RG, Jauch EC, Kern KB, Laurent I, Longstreth WT, Merchant RM, Morley P, Morrison LJ, Nadkarni V, Peberdy MA, Rivers EP, Rodriguez-Nunez A, Sellke FW, Spaulding C, Sunde K, Hoek TV. Post-cardiac arrest syndrome: epidemiology, pathophysiology, treatment, and prognostication. A Scientific Statement from the International Liaison Committee on Resuscitation; the American Heart Association Emergency Cardiovascular Care Committee; the Council on Cardiovascular Surgery and Anesthesia; the Council on Cardiopulmonary, Perioperative, and Critical Care; the Council on Clinical Cardiology; the Council on Stroke. Resuscitation. 2008 Dec;79(3):350-79. doi: 10.1016/j.resuscitation.2008.09.017. Epub 2008 Oct 28. PMID 18963350
- [Result] Mentzelopoulos SD, Zakynthinos SG. Post-cardiac arrest syndrome: pathological processes, biomarkers and vasopressor support, and potential therapeutic targets. Resuscitation. 2017 Dec;121:A12-A14. doi: 10.1016/j.resuscitation.2017.10.013. Epub 2017 Oct 18. No abstract available. PMID 29055751
- [Result] Zheng J, Lv C, Zheng W, Zhang G, Tan H, Ma Y, Zhu Y, Li C, Han X, Yan S, Pan C, Zhang J, Hou Y, Wang C, Bian Y, Liu R, Cheng K, Ma J, Zheng Z, Song R, Wang M, Gu J, McNally B, Ong MEH, Chen Y, Xu F; BASIC-OHCA Coordinators and Investigators. Incidence, process of care, and outcomes of out-of-hospital cardiac arrest in China: a prospective study of the BASIC-OHCA registry. Lancet Public Health. 2023 Dec;8(12):e923-e932. doi: 10.1016/S2468-2667(23)00173-1. Epub 2023 Sep 16. PMID 37722403